CLINICAL TRIAL: NCT03105544
Title: Improving Detection of Fetuses at Risk - Who Needs Systematic Training?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Lisbeth Andreasen, MD, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OBSTSIM
Record Dates: First submitted 2017-01-30; First posted 2017-04-10 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Improving Obstetric Ultrasound Skills
Keywords: simulation-based training; obstetric ultrasound; intrauterine growth restriction; ultrasound simulation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Simulation-based training: Virtual-reality simulation training on the Medaphor Scantrainer Transabdominal Simulator until expert level is reached. Then training on a physical mannikin until an average OSAUS-score of 3 or more is attained.
  Interventions: Other: simulation-based training
- Control (No Intervention): No intervention.

INTERVENTIONS:
Other: simulation-based training — As described under group descriptions
  Arms: Intervention

SUMMARY:
Detection of growth restricted fetuses relies primarily on abdominal ultrasound examinations during pregnancy. Many clinicians, however, have not received systematic training and may therefore perform inadequately. We wish to examine, whether systematic, simulation-based training can improve diagnostic accuracy of estimated fetal weight by ultrasound at different levels of clinical experience.

DETAILED DESCRIPTION:
Participants are physicians working at obstetric departments. Participant characteristics (age, experience in years and number of monthly scans) are recorded. Participants perform two abdominal growth scans prior to randomization and estimated fetal weight is compared to birth weight. Mean absolute percentage error is calculated as a measure of diagnostic accuracy.

Participants are then randomized to either control (no intervention) or intervention. The latter group receives training on the Metaphor Scantrainer trans abdominal ultrasound simulator until they pass a previously validated test. After completing the training the participants use a mannikin to practice systematic approach and 'knobology'.

All participants then perform another two growth scans. Diagnostic accuracy before and after the intervention or control period is compared.

We wish to examine the effect of systematic training on the diagnostic accuracy of estimated fetal weight by ultrasound across different levels of clinical experience.

If an effect can be found in the inexperienced participants, simulation-based training in obstetric ultrasound could be implemented as a part of basic obstetric training and/or as a means of maintaining skills.

ELIGIBILITY:
Inclusion Criteria:

* proficiency in the Danish language
* no prior experience with obstetric ultrasound simulation
* doctors who work within the field of gynecology and obstetrics

Exclusion Criteria:

* lack of proficiency in the Danish language
* prior experience with obstetric ultrasound simulation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of estimated fetal weight by ultrasound. | 1 month
  percentage error of fell weight estimate compared to actual fetal weight

SECONDARY OUTCOMES:
Ratings of ultrasound images | 1 month
  Images are rated using the image-scoring method by Salomon et al. (Salomon et al. Feasibility and reproducibility of an image-scoring method for quality control of fetal biometry in the second trimester. Ultrasound Obstet Gynecol 2006;27;34-40) The images are scores on the number of landmarks, correct caliper placement and image optimization. A minimum of 0 and a maximum of 16 points can be given (best possible score).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Tabor, DMSc, Study Director — Copenhagen University Hospital at Herlev
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen
  - Departments of Gynecology and Obstetrics, Hillerød Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Undecided